CLINICAL TRIAL: NCT03039764
Title: The Comparison Study of Virtual Reality Rehabilitation With Standard Occupational Therapy Versus Standard Occupational Therapy
Brief Title: Effects of Virtual Reality Based Rehabilitation in Acute Stroke Patients in an Inpatient Rehab Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Paused due to COVID and the study has expired. The PI left the institution in 2021 and another PI has not been assigned.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-6572
Record Dates: First submitted 2017-01-17; First posted 2017-02-01 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Stroke Syndrome; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard occupational therapy (No Intervention): This group will receiving standard occupational therapy for the treatment of acute stroke.
- SOT plus VR Rapael (Experimental): This group will receive virtual reality-based rehabilitation intervention wearing Rapael glove made by Neofect supplemented with standard occupational services per conventional protocols.
  Interventions: Device: Rapael

INTERVENTIONS:
Device: Rapael — This group will receive virtual reality-based rehabilitation intervention wearing Rapael glove made by Neofect supplemented with standard occupational services per conventional protocols.
  Arms: SOT plus VR Rapael

SUMMARY:
To evaluate the effects of virtual reality-based rehabilitation (Neofect Glove) for newly diagnosed cognitively intact adult dominant hemisphere stroke patients with paresis of their hand in supplementation with conventional occupational therapy to assess whether it improves motor function and speed recovery during inpatient rehabilitation versus conventional occupational therapy alone. Also, what impact does this have on quality of life.

DETAILED DESCRIPTION:
The American Stroke Association states that stroke is 5th leading cause of death in the United States and one of the leading causes of disability and loss of motor function. Approximately 80% of stroke survivors have upper extremity limitations where the distal upper extremity motor function is severely affected and is the last body part to recover. Restoration of arm function is essential to regaining activities of daily living (ADL) such as holding objects like utensils, turning a doorknob, writing or telephone use. Literature search shows that intensive and repetitive training may be necessary to modify neural organization and recover functional motor skills. Along with traditional rehabilitation methods, virtual reality (VR) based rehabilitation has emerged in recent years. VR-based rehabilitation is more intensive, of longer duration and more repetitive. Using VR rehabilitation, repetitive dull exercises can turn into a more challenging and motivating tasks such as games. Moreover, VR-based rehabilitation can provide a quantitative measure of the rehabilitation progress.

The investigators propose a study comparing conventional occupational services versus virtual reality-based rehabilitation intervention for participants during acute phase of stroke in the inpatient rehabilitation setting. The investigators hypothesize that by using VRA, will see a significant increase in the overall motor function, shorter hospital course and improved quality of life for the participants.

ELIGIBILITY:
Inclusion Criteria

* Minimum age of 18 years' old
* Unilateral upper extremity functional deficits after stroke
* First ever clinical diagnosis of stroke in the dominant hemisphere
* Diagnosis of ischemic or hemorrhagic stroke with unilateral paresis of dominant hand

Exclusion Criteria:

* Age less than 18 years' old
* Cognitive impairment resulting in inability to participate
* Severe aphasia resulting in inability to communicate to give consent or participate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with occupational therapy and with VR device will be assesed by Wolf Motor Function Test | 3 Months
  Scores on the Wolf Motor Function test measured at baseline and after therapy will be summarized using standard descriptive statistics for each treatment group. Data will be collected by designated research fellow.

SECONDARY OUTCOMES:
Number of participants treated with occupational therapy and with VR device will be assesed by Michigan Hand Outcome Questionnaire | 3 Months
  Scores of Michigan Hand Outcome Questionnaire measured at baseline and after therapy will be summarized using standard descriptive statistics for each treatment group. Data will be collected by designated research fellow.

CONTACTS AND LOCATIONS:
Locations (1):
- Burke rehabilitation Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
Will not share IPD